CLINICAL TRIAL: NCT06917976
Title: Evaluating the Effects of Psychological Stress on Salivary Biomarkers in Pediatric Patients
Brief Title: Evaluating the Effects of Psychological Stress on Salivary Biomarkers in Pediatric Patients Visiting Pediatric and General Dental Clinic
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Donya ali abd alkadim, master student, Al-Mustansiriyah University
Other Study IDs: AL- Mustansiriyah University
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Salivary Cortisol; Salivary Alpha Amylase

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: to compare the effect of environment and attitude of dentist in children visiting specialized pediatric dental clinic and general dental clinic . — the investigators will measure salivary cortisol and salivary alpha amylase and using children fear dental survey schedule - dental subscale

SUMMARY:
the goal of this study is to test the effect of psychological stress on pediatric patients visiting specialized and general dental clinic by measure salivary cortisol and salivary alpha amylase and by use children fear survey schedule -dental subscale .

80 male subjects will be enrolled in this study between 4-6 years old with first dental visit ,40 subjects visiting specialized pediatric dental clinic to see the effect of specific environment and attitude of dentist on child stress ,and 40 subjects visiting general dental clinic with normal environment and general dentist .

the method of study is by taking two saliva sample from child , first when he will enter the clinic at reception and second after half hour when he will diagnosed without any type of treatment.

ELIGIBILITY:
Inclusion Criteria:

* male
* 4-6 years old
* first dental visit
* patients with no systemic disease

Exclusion Criteria:

* medically compressed patient
* patients with systemic disease

Ages: 4 Years to 6 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: male children from 4-6 years old with first dental clinic
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
salivary alpha amylase | Baseline: saliva collection for cortisol and salivary alpha amylase measurement. up to half hour :saliva collection will be performed again as described at base line visit.
  measure salivary alpha amylase before and after half hour to see if the environment and attitude of dentist effect on salivary alpha amylase hormone.
salivary cortisol | Baseline: saliva collection for cortisol and salivary alpha amylase measurement. up to half hour :saliva collection will be performed again as described at base line visit.
  measure salivary cortisol before and after half hour to see if the environment and attitude of dentist effect on cortisol hormone.

IPD SHARING:
Plan to Share IPD: No